CLINICAL TRIAL: NCT05869149
Title: Systems Science Approaches to Improve Access to Healthier Foods: The FRESH Trial
Acronym: FRESH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: George Washington University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01MD018022-02 (NIH); IRB00024491 (Other: JHSPH IRB)
Record Dates: First submitted 2023-05-09; First posted 2023-05-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy Eating Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restaurants receiving FRESH intervention (Experimental): Restaurants enrolled in the experimental arm of will FRESH undergo activities aimed to improve their healthy food offerings at their restaurants.
  Interventions: Behavioral: Multilevel restaurant intervention to improve the food environment
- Restaurants not receiving FRESH intervention (No Intervention): Restaurants will be enrolled in the study, but not receive the FRESH intervention.

INTERVENTIONS:
Behavioral: Multilevel restaurant intervention to improve the food environment — FRESH is a restaurant-based intervention in low-income neighborhoods in Baltimore, MD and the Washington, District of Columbia metro area that aims to improve the healthy prepared-food environment for consumers, informed by community members and other stakeholders. FRESH intervention components include food preparation, food access and procurement, and consumer nutrition environment. Activities will take place over 16 months, and include training restaurant chefs to use healthier cooking methods, partnering with restaurant suppliers to offer healthier ingredients, and offering point-of-purchase promotions to educate customers on the healthier promoted food options. Intervention staff will form strong relationships with restaurant owners and chefs via in-person visits at least twice a month. Data from the intervention trial will inform the development of a system dynamics simulation model that will allow stakeholders to test new policy ideas prior to implementation.
  Arms: Restaurants receiving FRESH intervention

SUMMARY:
Working with independently owned restaurants, a common source of calorie-rich, nutrient-poor foods in predominantly minority, low-income urban neighborhoods, has the potential to improve dietary quality, and contribute to cancer prevention. This study uses systems science approaches to improve access to healthier foods in independently owned restaurants by: 1) testing the effects of a novel intervention called FRESH (Focus on Restaurant Engagement to Strengthen Health) on dietary quality, health indicators and other outcomes in African American and Latin communities, and 2) developing a system dynamics model to allow stakeholders to virtually test FRESH strategies in their own communities. The resulting restaurant intervention simulation model offers potential cost savings from avoided trial-and-error testing, and will support community-based cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-75 years)
* Regular restaurant customer (e.g., visits the specified restaurant at least 1x/week)
* Live in a household of at least 2 persons (criterion intended to provide a more stable sample, and to reduce loss to follow-up)
* Current resident of study neighborhood

Exclusion Criteria:

* Anticipate moving out of Baltimore or District of Columbia metropolitan area in the next 18 months
* Pregnant (due to changes in diet, weight and body composition)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Customer Dietary Quality | 1 hour, 24 months apart
  Regular customer diet quality in the last 30 days will be assessed using the 2014 semi-quantitative Block Food Frequency Questionnaire (FFQ). The FFQ provides the data that allows for calculating the Healthy Eating Index. We will use the 2015 index rules. Healthy Eating Index (HEI) 2015 Score and individual component scores will be calculated from the FFQ according to the HEI-2015 guidelines to assess changes in overall diet quality and changes within each component. The range of scores for the Healthy Eating Index 2015 is 0-100. A higher score is considered better and represents meeting more of the recommended dietary guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Gittlesohn, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colon-Ramos U, Lewis EC, Tucker AC, Poirier L, Pathiravasan CH, Estrade M, Igusa T, Wolfson JA, Mui Y, Velez-Burgess V, Thomas AE, Hua S, Cheskin LJ, Trujillo AJ, Oladimeji AT, Williamson S, Romero R, Hernandez PS, Gittelsohn J. Design of the Focus on Restaurant Engagement to Strengthen Health (FRESH) study: leveraging systems science to work with independently-owned restaurants to increase access to and promotion of healthful foods. Front Public Health. 2025 Jan 7;12:1427792. doi: 10.3389/fpubh.2024.1427792. eCollection 2024. PMID 39845656